CLINICAL TRIAL: NCT04403269
Title: "STUDY OF THE EFFICIENCY OF NORMAL HUMAN IMMUNOGLOBULINS (IVIG) IN PATIENTS AGED 75 YEARS AND OVER COVID-19 WITH SEVERE ACUTE RESPIRATORY FAILURE" GERONIMO 19
Brief Title: NORMAL HUMAN IMMUNOGLOBULINS (IVIG) IN PATIENTS AGED 75 YEARS AND OVER, COVID-19 WITH SEVERE ACUTE RESPIRATORY FAILURE
Acronym: GERONIMO 19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Dr Laure PARNET, Principal Investigator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P20/07 GERONIMO 19
Record Dates: First submitted 2020-05-18; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Sars-CoV2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IgIV (Experimental): The experimental arm is human immunoglobulins. 2 infusion at D1 and D2. (0.8 g / kg by IV infusion)
  Interventions: Drug: IgIV

INTERVENTIONS:
Drug: IgIV — 2 infusion at D1 and D2 (0.8 g / kg by IV infusion)

SUMMARY:
According to recent data, death rate is more than 20% for 75 years old hospitalized patients and older.

In case of aggravation, according to the latest observations, if they are refused for mechanical ventilation in intensive care, their death rate could reach 60% even for patients without comorbidity.

Apart from an increase in oxygen therapy, no specific treatment is currently proposed.

The control of the inflammatory component seems to be a key element to be able to influence the patients' health evolution.

Polyvalent intravenous immunoglobilins have immunomodulatory and anti-inflammatory properties with a favorable safety profile for these elderly patients and several clinical cases lead to positive impact in the caring for Covid patients.

This study objective is evaluation of the efficacy of polyvalent IVIg in combination with the standard management of patients aged 75 and over with SARSCov2 infection with acute respiratory failure (saturation ≤ 95%) requiring oxygen therapy> 5 L / min (i.e. patients considered as moderate to severe ARDS according to the Berlin definition, Pa02 / Fi02≤200) and disqualified from a care in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged 75 and over
* SARS-coV2 infection confirmed by RT-PCR or thoraco-pulmonary CT
* Hospitalized in the acute general geriatrics unit of the Versailles Hospital Center
* Patient rejected from resuscitation
* Saturation ≤ 95% under oxygen therapy> 5 L / min (i.e. PaO2 / FiO2≤200mmHg according to the Berlin definition of ARDS) by means of a nasal cannula, a high concentration facial mask or another device similar oxygen distribution

Exclusion Criteria:

* Patient under palliative care
* Patient with contraindication to IV polyvalent Ig

  1. . Hypersensitivity to the active substance or to any of the excipients (L-proline)
  2. . Hypersensitivity to human immunoglobulins, especially when the patient has anti-IgA antibodies,
  3. . Patients with type I or II hyperprolinemia
* Patient under guardianship or curatorship
* Patient receiving another experimental treatment as part of an interventional study
* Moderate to severe dementia known: it must have been diagnosed before hospitalization and is defined by an MMSE <20/30 or a neuropsychological assessment with a diagnosis made.
* Patient not affiliated with a social security system in France
* ADL patients <4/6 and / or IADL <6/8

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-05-05 (Estimated); Study Completion 2021-05-05 (Estimated)

PRIMARY OUTCOMES:
Mortality | Day 14

SECONDARY OUTCOMES:
Total number of days of full hospitalization | 3 and 6 months
Duration of oxygen therapy | 3 and 6 months
Ferritin level in the blood | 3 and 6 months
CRP level in the blood | 3 and 6 months
LDH level in the blood | 3 and 6 months
Lymphocyte level in the blood | 3 and 6 months
PNN level in the blood | 3 and 6 months
platelet level in the blood | 3 and 6 months
WHO performance index | 3 and 6 months
WHOQOL-OLD questionnaire | 3 and 6 months
Lung function by pulmonary computed tomography | 3 and 6 months
Lung function by EFR | 3 and 6 months
Mortality | 3 and 6 months
Readmission Rates | 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Versailles, Le Chesnay, France